CLINICAL TRIAL: NCT01013831
Title: A Phase I Study of Erlotinib in Patients With Premalignant Lesions of the Lung
Brief Title: Erlotinib Hydrochloride in Preventing Cancer in Patients With Precancerous Lesions of the Lung
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NCI-2013-00750; NCI-2013-00750 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); RPCI-I-121507; NU-NWU08-11-01; STU00012618; NCI 08-11-01 (Other: Northwestern University); NWU08-11-01 (Other: DCP); P30CA060553 (NIH); N01CN35157 (NIH)
Record Dates: First submitted 2009-11-13; First posted 2009-11-16 (Estimated); Last update posted 2015-02-18 (Estimated); Status verified 2014-04

CONDITIONS: Dysplasia; Metaplasia; Pulmonary Precancerous Condition
MeSH Terms: conditions — Metaplasia | interventions — Erlotinib Hydrochloride

ARMS (1):
- Prevention (erlotinib hydrochloride) (Experimental): Patients receive erlotinib hydrochloride PO QD for 90 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Erlotinib Hydrochloride; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study

INTERVENTIONS:
Drug: Erlotinib Hydrochloride — Given PO
  Other Names: Cp-358,774
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
This phase I trial studies the side effects and best dose of erlotinib hydrochloride in preventing cancer in patients with precancerous lesions of the lung. Erlotinib hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the lowest dose of erlotinib (erlotinib hydrochloride) that will decrease the ratio of phosphorylated to total epidermal growth factor receptor (EGFR) (phosphorylated EGFR [pEGFR]/EGFR) by at least 20% in subjects with premalignant lesions of the lung. This will be accomplished by implementing a dose de-escalation trial of erlotinib (i.e., 75, 50, and 25 or 100 mg by mouth daily for a 3-month period), and determining the pEGFR/EGFR ratio in premalignant lesions of the lung epithelium by immunohistochemistry. Changes in the pEGFR/EGFR ratio will be assessed by comparing the pre-treatment (baseline) ratio to that of the post-treatment (3 month) ratio, measured in paraffin embedded biopsy specimens.

SECONDARY OBJECTIVES:

I. To determine the effect of erlotinib on the following biomarkers of potential biological relevance in paraffin embedded lung biopsies, p-v-akt murine thymoma viral oncogene homolog 1 (Akt), p-mitogen-activated protein kinase 1 (Erk), and marker of proliferation Ki-67 (Ki67).

II. To characterize the toxicity profile of erlotinib in this cohort of subjects.

III. To analyze and model erlotinib's pharmacokinetic/pharmacodynamic (PK/PD) profile. Serial blood samples will be drawn at the beginning and at the end of erlotinib treatment, and pharmacokinetic parameters will be determined. The status of EGFR genotype (and that of others genes linked to erlotinib PK/PD) clinical toxicity, and dose will be examined as possible other influential covariates by comparing them to experimentally measured PK profiles, and PD profiles (in particular, the pEGFR/EGFR ratio). The goal of these studies will be to determine the optimal biologic concentration (OBC) of Erlotinib that is associated with the lowest toxicity and highest effect, for a given subject's pharmacogenomic profile.

OUTLINE:

Patients receive erlotinib hydrochloride orally (PO) once daily (QD) for 90 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a premalignant lung lesion (metaplasia or dysplasia) on autofluorescent bronchoscopy (AFB) within 1 month
* Participants must have a >= 10 pack year lifetime smoking history; current and former smokers only are eligible for this trial
* No contraindications for treatment with erlotinib or additional bronchoscopies
* Absolute neutrophil count (ANC) of >= 1.5 x 10^9/L
* Platelet count of >= 100 x 10^9/L
* Creatinine level of less than 1.5 mg/dL
* Total bilirubin =< 2.0 mg/dl
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 1.5 x upper limit of normal (ULN)
* Alkaline phosphatase =< 2.5 x ULN
* Must meet Eastern Cooperative Oncology Group (ECOG) performance status criteria of 0-1
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) throughout the duration of the study and for 1 month following cessation of study drug; females must begin adequate contraception immediately following screening pregnancy test; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her study physician immediately; if she is pregnant, she will be immediately withdrawn from the study
* Ability to understand and the willingness to sign a written institutional review board (IRB) approved informed consent document

Exclusion Criteria:

* Subjects with life-threatening medical conditions that would preclude the treatment intervention and bronchoscopy, including, but not limited to, unstable pulmonary function, acute cardiac failure, which is unstable despite medication use; uncontrolled hypertension; uncontrolled diabetes mellitus; unstable coronary artery disease; acute or chronic liver disease, ongoing or active infection; or psychiatric illness/social situations that would limit compliance with study requirements
* Participants with evidence of an active cancer or carcinoma in situ, are not eligible
* Participants currently taking medications that induce or inhibit the cytochrome P450, family 3, subfamily A, polypeptide 4-7 (CYP3A4-7) enzymes
* Participants may not be receiving any other investigational agents within 3 months
* Participants taking warfarin
* History of allergic reactions attributed to erlotinib, a known hypersensitivity to erlotinib, or agents with a similar chemical or biological composition to erlotinib
* Women who are pregnant or lactating are excluded from the study because based on the proposed mechanism of tyrosine kinase inhibition of erlotinib; erlotinib should be assumed to cause fetal harm when administered to a pregnant woman; there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with erlotinib
* History of interstitial lung disease (ILD)

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-10; Primary Completion 2012-02 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Change in the ratio of p-EGFR to total EGFR | Baseline up to 90 days

SECONDARY OUTCOMES:
Change in the expression of p-Akt | Baseline up to 90 days
  Analyzed using an analysis-of-variance (ANOVA) on the change from baseline expression level with a factor for dose (75, 50, 25 or 100). All tests will be two-sided and tested at level alpha=0.05. If the overall comparison is significant, pairwise comparisons will be done using straight Bonferroni adjustments.
Change in the expression of p-Erk | Baseline up to 90 days
  Analyzed using an ANOVA on the change from baseline expression level with a factor for dose (75, 50, 25 or 100). All tests will be two-sided and tested at level alpha=0.05. If the overall comparison is significant, pairwise comparisons will be done using straight Bonferroni adjustments.
Change in the expression of Ki67 | Baseline up to 90 days
  Analyzed using an ANOVA on the change from baseline expression level with a factor for dose (75, 50, 25 or 100). All tests will be two-sided and tested at level alpha=0.05. If the overall comparison is significant, pairwise comparisons will be done using straight Bonferroni adjustments.
Incidence of toxicities, graded according to Common Toxicity Criteria, version 3.0 | Up to 30 days

OTHER OUTCOMES:
PK/PD parameters | Up to 90 days
Pharmacogenomic profile | Up to 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Seema Khan, Principal Investigator — Northwestern University
Locations (4):
- United States (4):
  - Northwestern University, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Boston University School of Medicine, Boston, Massachusetts
  - Roswell Park Cancer Institute, Buffalo, New York